CLINICAL TRIAL: NCT03213678
Title: NCI-COG Pediatric MATCH (Molecular Analysis For Therapy Choice)- Phase 2 Subprotocol of LY3023414 in Patients With Solid Tumors
Brief Title: Samotolisib in Treating Patients With Relapsed or Refractory Advanced Solid Tumors, Non-Hodgkin Lymphoma, or Histiocytic Disorders With TSC or PI3K/MTOR Mutations (A Pediatric MATCH Treatment Trial)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-01249; NCI-2017-01249 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); APEC1621D; APEC1621D (Other: Children's Oncology Group); APEC1621D (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2017-07-10; First posted 2017-07-11 (Actual); Results first posted 2024-09-04 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Advanced Malignant Solid Neoplasm; Ann Arbor Stage III Non-Hodgkin Lymphoma; Ann Arbor Stage IV Non-Hodgkin Lymphoma; Malignant Glioma; Recurrent Ependymoma; Recurrent Ewing Sarcoma; Recurrent Glioma; Recurrent Hepatoblastoma; Recurrent Langerhans Cell Histiocytosis; Recurrent Malignant Germ Cell Tumor; Recurrent Malignant Solid Neoplasm; Recurrent Medulloblastoma; Recurrent Neuroblastoma; Recurrent Non-Hodgkin Lymphoma; Recurrent Osteosarcoma; Recurrent Peripheral Primitive Neuroectodermal Tumor; Recurrent Primary Central Nervous System Neoplasm; Recurrent Rhabdomyosarcoma; Recurrent Soft Tissue Sarcoma; Refractory Langerhans Cell Histiocytosis; Refractory Malignant Germ Cell Tumor; Refractory Malignant Solid Neoplasm; Refractory Neuroblastoma; Refractory Non-Hodgkin Lymphoma; Refractory Primary Central Nervous System Neoplasm; Rhabdoid Tumor; Stage III Osteosarcoma AJCC v7; Stage III Soft Tissue Sarcoma AJCC v7; Stage IV Osteosarcoma AJCC v7; Stage IV Soft Tissue Sarcoma AJCC v7; Stage IVA Osteosarcoma AJCC v7; Stage IVB Osteosarcoma AJCC v7; Wilms Tumor
MeSH Terms: conditions — Glioma; Ependymoma; Sarcoma, Ewing; Hepatoblastoma; Histiocytosis, Langerhans-Cell; Medulloblastoma; Neuroblastoma; Lymphoma, Non-Hodgkin; Osteosarcoma; Neuroectodermal Tumors, Primitive, Peripheral; Central Nervous System Neoplasms; Rhabdomyosarcoma; Sarcoma; Rhabdoid Tumor; Wilms Tumor | interventions — Specimen Handling; Magnetic Resonance Spectroscopy; LY3023414; X-Rays; Phantoms, Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (samotolisib) (Experimental): Patients receive samotolisib PO BID on days 1-28. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unexpected toxicity. Patients undergo an x-ray, CT, MRI, FDG-PET, and blood sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: FDG-Positron Emission Tomography; Procedure: Magnetic Resonance Imaging; Drug: Samotolisib; Procedure: X-Ray Imaging

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood specimen collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: FDG-Positron Emission Tomography — Undergo FDG-PET
  Other Names: FDG; FDG-PET; FDG-PET Imaging
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Samotolisib — Given PO
  Other Names: 2H-Imidazo(4,5-C)quinolin-2-one, 1,3-Dihydro-8-(5-(1-hydroxy-1-methylethyl)-3-pyridinyl)-1-((2S)-2-methoxypropyl)-3-methyl-; LY 3023414; LY-3023414; LY3023414; WHO 10889
Procedure: X-Ray Imaging — Undergo x-ray
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiographic imaging procedure (procedure); Radiography; RG; Static X-Ray; X-Ray

SUMMARY:
This phase II Pediatric MATCH trial studies how well samotolisib works in treating patients with solid tumors, non-Hodgkin lymphoma, or histiocytic disorders with TSC or PI3K/MTOR mutations that have spread to other places in the body (metastatic) and have come back (recurrent) or do not respond to treatment (refractory). Samotolisib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the objective response rate (ORR; complete response + partial response) in pediatric patients treated with samotolisib (LY3023414) with advanced solid tumors, non-Hodgkin lymphomas or central nervous system (CNS) tumors that harbor TSC loss of function mutations, and/or other PI3K/MTOR activating mutations.

SECONDARY OBJECTIVES:

I. To estimate the progression free survival in pediatric patients treated with LY3023414 with advanced solid tumors, non-Hodgkin lymphomas or CNS tumors that harbor TSC loss of function mutations, and/or other PI3K/MTOR activating mutations.

II. To obtain information about the tolerability of LY3023414 in children with relapsed or refractory cancer.

III. To characterize the pharmacokinetics of LY3023414 in children with recurrent or refractory cancer.

EXPLORATORY OBJECTIVES:

I. To increase knowledge of the genomic landscape of relapsed pediatric solid tumors and lymphomas and identify potential predictive biomarkers (other than the genomic alteration for which study treatment was assigned) using additional genomic, transcriptomic, and proteomic testing platforms.

II. To explore approaches to profiling changes in tumor genomics over time through evaluation of circulating tumor deoxyribonucleic acid (DNA).

III. To evaluate the frequency and mechanism of biallelic loss of function, and evaluate the expression of TSC1, TSC2, and PTEN in subjects who enroll with a loss of function mutation in one of these genes.

OUTLINE: This is a dose-escalation study.

Patients receive samotolisib orally (PO) twice daily (BID) on days 1-28. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unexpected toxicity. Patients undergo an x-ray, computed tomography (CT), magnetic resonance imaging (MRI), fludeoxyglucose F-18 (FDG)-position emission tomography (FDG-PET), and blood sample collection on study.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have enrolled onto APEC1621SC/NCI-2017-01251/ NCT03155620 and must have been given a treatment assignment to Molecular Analysis for Therapy Choice (MATCH) to APEC1621D based on the presence of an actionable mutation as defined in APEC1621SC; note that treatment assignment may be to primary cohort A for patients with TSC1 or TSC2 loss of function mutations or primary cohort B for patients with other PI3K/MTOR pathway mutations
* Patients accruing to dose level 1 must have a body surface area >= 0.52 m^2 at the time of study enrollment; patients accruing to dose level 2 must have a body surface area >= 0.37 m^2 at the time of study enrollment; patients accruing to dose level -1 must have a body surface area >= 0.75 m^2 at the time of study enrollment
* Patients must have radiographically measurable disease at the time of study enrollment; patients with neuroblastoma who do not have measurable disease but have metaiodobenzylguanidine (MIBG) positive (+) evaluable disease are eligible; measurable disease in patients with CNS involvement is defined as any lesion that is at minimum 10 mm in one dimension on standard magnetic resonance imaging (MRI) or computed tomography (CT)

  * Note: The following do not qualify as measurable disease:

    * Malignant fluid collections (e.g., ascites, pleural effusions)
    * Bone marrow infiltration except that detected by MIBG scan for neuroblastoma
    * Lesions only detected by nuclear medicine studies (e.g., bone, gallium or positron emission tomography [PET] scans) except as noted for neuroblastoma
    * Elevated tumor markers in plasma or cerebrospinal fluid (CSF)
    * Previously radiated lesions that have not demonstrated clear progression post radiation
    * Leptomeningeal lesions that do not meet the measurement requirements for Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
    * Bone lesions without an associated soft tissue mass >= 10 mm in greatest diameter; bone lesions with an associated soft tissue mass >= 10 mm in greatest diameter imaged by CT or MRI are considered measurable
* Karnofsky >= 50% for patients > 16 years of age and Lansky >= 50 for patients =< 16 years of age; Note: neurologic deficits in patients with CNS tumors must have been stable for at least 7 days prior to study enrollment; patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Patients must have fully recovered from the acute toxic effects of all prior anti-cancer therapy and must meet the following minimum duration from prior anti-cancer directed therapy prior to enrollment; if after the required timeframe, the numerical eligibility criteria are met, e.g. blood count criteria, the patient is considered to have recovered adequately

  * Cytotoxic chemotherapy or other anti-cancer agents known to be myelosuppressive; >= 21 days after the last dose of cytotoxic or myelosuppressive chemotherapy (42 days if prior nitrosourea)
  * Anti-cancer agents not known to be myelosuppressive (e.g. not associated with reduced platelet or absolute neutrophil count [ANC] counts): >= 7 days after the last dose of agent
  * Antibodies: >= 21 days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to grade =< 1
  * Corticosteroids: if used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid
  * Hematopoietic growth factors: >= 14 days after the last dose of a long-acting growth factor (e.g. pegfilgrastim) or 7 days for short-acting growth factor; for growth factors that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur; the duration of this interval must be discussed with the study chair and the study-assigned research coordinator
  * Interleukins, interferons and cytokines (other than hematopoietic growth factors): >= 21 days after the completion of interleukins, interferon or cytokines (other than hematopoietic growth factors)
  * Stem cell Infusions (with or without total body irradiation [TBI]):

    * Allogeneic (non-autologous) bone marrow or stem cell transplant, or any stem cell infusion including donor lymphocyte infusion (DLI) or boost infusion: >= 84 days after infusion and no evidence of graft versus host disease (GVHD)
    * Autologous stem cell infusion including boost infusion: >= 42 days
  * Cellular therapy: >= 42 days after the completion of any type of cellular therapy (e.g. modified T cells, natural killer [NK] cells, dendritic cells, etc.)
  * Radiation therapy (XRT)/external beam irradiation including protons: >= 14 days after local XRT; >= 150 days after TBI, craniospinal XRT or if radiation to >= 50% of the pelvis; >= 42 days if other substantial bone marrow (BM) radiation

    * Note: radiation may not be delivered to "measurable disease" tumor site(s) being used to follow response to subprotocol treatment
  * Radiopharmaceutical therapy (e.g., radiolabeled antibody, iobenguane I-131 [131I-MIBG]): >= 42 days after systemically administered radiopharmaceutical therapy
  * Patients must not have received prior exposure to LY3023414
  * Patients must not have received prior exposure to an agent specifically directed at the PI3K/MTOR pathway (a PI3K inhibitor, an AKT inhibitor, an MTOR inhibitor, including rapalogs, or a combined PI3K/MTOR inhibitor)
* For patients with solid tumors without known bone marrow involvement:

  * Peripheral absolute neutrophil count (ANC) >= 1000/mm^3
  * Platelet count >= 100,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
* Patients with known bone marrow metastatic disease will be eligible for study provided they meet the blood counts (may receive transfusions provided they are not known to be refractory to red cell or platelet transfusions); these patients will not be evaluable for hematologic toxicity
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 ml/min/1.73 m^2 or a serum creatinine based on age/gender as follows:

  * Age: 1 to < 2 years; maximum serum creatinine (mg/dL): male 0.6; female 0.6
  * Age: 2 to < 6 years; maximum serum creatinine (mg/dL): male 0.8; female 0.8
  * Age: 6 to < 10 years; maximum serum creatinine (mg/dL): male 1; female 1
  * Age: 10 to < 13 years; maximum serum creatinine (mg/dL): male 1.2; female 1.2
  * Age: 13 to < 16 years; maximum serum creatinine (mg/dL): male 1.5; female 1.4
  * Age: >= 16 years; maximum serum creatinine (mg/dL): male 1.7; female 1.4
* Bilirubin (sum of conjugated + unconjugated) =< 1.5 x upper limit of normal (ULN) for age
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 135 U/L; (for the purpose of this study, the ULN for SGPT is 45 U/L)
* Serum albumin >= 2 g/dL
* Patients must have a normal blood sugar level for age; if an initial random draw (i.e. non-fasting) blood glucose value is out of range, it is acceptable to repeat this test as a fasting draw
* Patients must have a serum triglyceride level =< 300 mg/dL and serum cholesterol level =< 300 mg/dL; if an initial random draw (i.e. non-fasting) is out of range, it is acceptable to repeat this test as a fasting draw
* Patients with seizure disorder may be enrolled if on anticonvulsants and well controlled
* Nervous system disorders (by Common Terminology Criteria for Adverse Events version 5.0 [CTCAE V 5.0]) resulting from prior therapy must be =< grade 2, with the exception of decreased tendon reflex (DTR); any grade of DTR is eligible
* Corrected QT (QTc) interval =< 480 milliseconds
* Patients must be able to swallow intact tablets
* All patients and/or their parents or legally authorized representatives must sign a written informed consent; assent, when appropriate, will be obtained according to institutional guidelines

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study; pregnancy tests must be obtained in girls who are post-menarchal; males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method while receiving study treatment and for 3 months after the last dose of LY3023414
* Concomitant medications

  * Corticosteroids: patients receiving corticosteroids who have not been on a stable or decreasing dose of corticosteroid for at least 7 days prior to enrollment are not eligible; if used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid
  * Investigational drugs: patients who are currently receiving another investigational drug are not eligible
  * Anti-cancer agents: patients who are currently receiving other anti-cancer agents are not eligible
  * Anti-GVHD agents post-transplant: patients who are receiving cyclosporine, tacrolimus or other agents to prevent graft-versus-host disease post bone marrow transplant are not eligible for this trial
* Patients who have an uncontrolled infection are not eligible
* Patients who have insulin dependent diabetes are not eligible
* Patients who have received a prior solid organ transplantation are not eligible
* Patients with subependymal giant cell astrocytomas (SEGAs) are not eligible
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible

Ages: 12 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theodore W Laetsch, Principal Investigator — Children's Oncology Group
Locations (127):
- United States (125):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Banner Children's at Desert, Mesa, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Puerto Rico (2):
  - San Jorge Children's Hospital, San Juan
  - University Pediatric Hospital, San Juan

REFERENCES:
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Samotolisib)
Started | 18
Completed | 0
Not Completed | 18
Not completed — Death | 1
Not completed — Physician Decision | 1
Not completed — Progressive disease | 16

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Samotolisib)
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.8 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 14
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: A responder is defined as a patient who achieves a best response of partial response or complete response on the study. Response rates will be calculated as the percent of evaluable patients who are responders. The revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) was used to determine response and progression in this study, with specific criteria outlined for the different subtypes of tumors (e.g., 2-dimensional measurements for central nervous system (CNS) tumors).
Time Frame: Up to 2 years from study entry
Population: One patient did not receive any protocol treatment and is excluded from this analysis.
Measure: Number (90% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (Samotolisib)
Number analyzed (Participants) | 17
percentage of patients | 0 [0 to 0]

2. Secondary Outcome: Percentage of Patients Experiencing Grade 3 or 4 Adverse Events
Description: Percentage of patients experiencing grade 3 or higher adverse events will be evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0
Time Frame: Up to 2 years from study entry
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Treatment (Samotolisib)
Number analyzed (Participants) | 17
Percentage of patients | 24 [7 to 50]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: The Kaplan-Meier method will be used to estimate the 3-month PFS. PFS is defined as time from initiation of protocol treatment to disease progression, recurrence, death from any cause, or date of last contact.
Time Frame: Up to 3 months from study entry
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Samotolisib)
Number analyzed (Participants) | 17
percentage of participants | 12 [2 to 31]

4. Secondary Outcome: Pharmacokinetic (PK) of Samotolisib, Area Under the Curve (AUC).
Description: The mean (sd) of the AUC
Time Frame: Up to day 15 of cycle 1
Population: Three of the enrolled patients had PK data available for analysis
Measure: Mean (Standard Deviation); unit: h*μg/mL
Arm/Group | Treatment (Samotolisib)
Number analyzed (Participants) | 3
h*μg/mL | 2323 (1006)

5. Other Pre Specified Outcome: Potential Predictive Biomarker Identification Using Additional Genomic, Transcriptomic, and Proteomic Testing Platforms
Description: A descriptive analysis will be performed and will be summarized with simple summary statistics. All of these analyses will be descriptive in nature.
Time Frame: Up to 3 years
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Biallelic Loss of Function Frequency and Mechanism
Description: as for outcome 5
Time Frame: Up to 3 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in Tumor Genomic Profile
Description: as for outcome 5
Time Frame: Baseline up to 3 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: TSC1, TSC2, and PTEN Expression Levels
Description: as for outcome 5
Time Frame: Up to 3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Events monitored/assessed from enrollment to 30 days after the end of treatment, up to 2 years. All-Cause Mortality monitored/assessed up to 5 years
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. All-Cause Mortality includes all deaths collected on the study. Ineligible patients are excluded from reporting of adverse events.
Arm/Group | Treatment (Samotolisib)
All-Cause Mortality (participants affected / at risk) | 14/18
Serious Adverse Events (participants affected / at risk) | 9/17
Other Adverse Events (participants affected / at risk) | 16/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Samotolisib) (N=17)
Heart failure (Cardiac disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Death NOS (General disorders) | 2
Disease progression (General disorders) | 1
Pain (General disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Lung infection (Infections and infestations) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Muscle weakness right-sided (Nervous system disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Samotolisib) (N=17)
Anemia (Blood and lymphatic system disorders) | 9
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 2
Endocrine disorders - Other, specify (Endocrine disorders) | 1
Blurred vision (Eye disorders) | 3
Dry eye (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Anal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 6
Diarrhea (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Esophagitis (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 9
Oral pain (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 5
Edema face (General disorders) | 1
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 11
Fever (General disorders) | 6
Gait disturbance (General disorders) | 1
Otitis media (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Bruising (Injury, poisoning and procedural complications) | 1
Activated partial thromboplastin time prolonged (Investigations) | 1
Alanine aminotransferase increased (Investigations) | 7
Alkaline phosphatase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 5
Blood bicarbonate decreased (Investigations) | 1
Blood bilirubin increased (Investigations) | 3
Blood lactate dehydrogenase increased (Investigations) | 1
CPK increased (Investigations) | 1
Cholesterol high (Investigations) | 3
Creatinine increased (Investigations) | 4
Lymphocyte count decreased (Investigations) | 7
Neutrophil count decreased (Investigations) | 4
Platelet count decreased (Investigations) | 4
Weight loss (Investigations) | 4
White blood cell decreased (Investigations) | 6
Anorexia (Metabolism and nutrition disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 8
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 2
Hyperphosphatemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 4
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 7
Hypophosphatemia (Metabolism and nutrition disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 6
Paresthesia (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 1
Irritability (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Urinary frequency (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Genital edema (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Laryngopharyngeal dysesthesia (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-28): https://cdn.clinicaltrials.gov/large-docs/78/NCT03213678/Prot_SAP_000.pdf